CLINICAL TRIAL: NCT00597714
Title: Efficacy Study of T Cell Depleted Allogeneic Non-myeloablative Stem Cell Transplantation
Brief Title: Efficacy Study of T Cell Depleted Allogeneic Non-myeloablative Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Rizzieri, MD (Other)
Responsible Party: Sponsor-Investigator, David Rizzieri, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00003567
Record Dates: First submitted 2008-01-14; First posted 2008-01-18 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-02

CONDITIONS: Hodgkin's Disease; Non Hodgkin's Lymphoma; Myeloma; Leukemia; Myelodysplasia
Keywords: Stem Cell Transplantation, Non-myeloablative
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Neoplasms, Plasma Cell; Leukemia; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A - Lymphoid Disease (Experimental): Group A: Patients with a high chance of progressive lymphoid or myelomatous disease undergo Non-myeloablative Stem Cell Transplantation.
  Interventions: Drug: Non-myeloablative Stem Cell Transplantation
- Cohort B - Myeloid Disease (Experimental): Group B: Patients with a high chance of progressive myeloid diseases, marrow failure syndromes or myeloproliferative disorders undergo Non-myeloablative Stem Cell Transplantation.
  Interventions: Drug: Non-myeloablative Stem Cell Transplantation
- Donor (No Intervention): Donor priming and apheresis will include filgrastim 8 mcg/kg subcutaneously twice daily for 4 days prior to stem cell collection and continuing until pheresis is completed. Alternative mobilization strategies may be employed at the investigator's discretion.

INTERVENTIONS:
Drug: Non-myeloablative Stem Cell Transplantation — The preparative regimen is 4 days of daily fludarabine at 40 mg/m2/d infused over 30 minutes; melphalan 140 mg/m2/d for 1 day administered over 15 minutes; 4 days of Alemtuzumab at 20 mg/d in 250 ml of normal saline infused over 3 hours. Group B's prep regimen will begin on day -5 or day -4 and busulfan 130mg/m2/d for 2 days over 3 hours. The peripheral blood stem cells (PBSCs) will be infused over 2-4 days. Patient evaluations will occur 2 times per week by physical exam for toxicity through day 45.
  Other Names: Allogeneic Stem Cell Transplant
  Arms: Cohort A - Lymphoid Disease; Cohort B - Myeloid Disease

SUMMARY:
The central hypothesis of this study is that use of a less toxic chemotherapy preparative regimen for allogeneic hematopoietic stem cell transplantation in combination with T cell depletion with alemtuzumab for patients with high risk hematologic malignancies will allow effective control of disease and improved disease free and overall survival compared with historical expectations. Specifically, the objectives are to estimate toxicity, disease free, progression free, event free, and overall survival rates in patients treated with alemtuzumab T cell depleted, reduced intensity preparative regimen followed by allogeneic hematopoietic transplantation; evaluate immune recovery following this reduced intensity allogeneic immunotherapy; develop an in vitro assay to allow patient individualized targeted dosing.

DETAILED DESCRIPTION:
The central hypothesis of this study is that use of a less toxic chemotherapy preparative regimen for allogeneic hematopoietic stem cell transplantation in combination with T cell depletion with alemtuzumab for patients with high risk hematologic malignancies will allow effective control of disease and improved disease free and overall survival compared with historical expectations. Specifically, the objectives are to estimate toxicity, disease free, progression free, event free and overall survival rates in patients treated with an alemtuzumab T cell depleted, reduced intensity preparative regimen followed by allogeneic hematopoietic transplantation; evaluate immune recovery following this reduced intensity allogeneic immunotherapy; develop an in vitro assay to allow patient individualized targeted dosing. The study population is HIV negative, adult patients who are not pregnant but have confirmed diagnosis of disease; must have Cancer and Leukemia Group B (CALGB) performance status (PS) 0, 1, or 2; must have a 3-6/6 human leukocyte antigen (HLA)-matched related donor or 8/8 (A, B, C, DRB1, DQ are the primary determinants) or better HLA-matched unrelated donor who is evaluated and deemed able to provide peripheral blood stem cells (PBPCs) and/or marrow by the transplant team. The target population of patients is those with a high chance of progressive lymphoid or myelomatous diseases, progressive myeloid diseases, marrow failure syndromes or myeloproliferative disorders.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Subjects must have their diagnosis confirmed at the transplant center.
* Performance status must be Cancer and Leukemia Group B (CALGB) = 0, 1, or 2.
* Subjects must have a 3-6/6 human leukocyte antigen (HLA)-matched related donor or 8/8 or better allele level match matched unrelated donor (MUD) (at A,B, C, DRB1, DQ).
* HIV negative.
* Women of child bearing potential must have a negative pregnancy test within 1 week of starting therapy.
* Subjects > or equal to 18 years of age are eligible.
* Subjects must have a Multi Gated Acquisition Scan (MUGA) and/or Echocardiography (ECHO) or cardiac magnetic resonance (MR) and or diffusing capacity testing of the lung for carbon monoxide (DLCO) performed before transplant.
* Specific populations:

  * Group A) Subjects with a high chance of progressive lymphoid or myelomatous diseases.
  * Group B) Subjects with a high chance of progressive myeloid diseases, marrow failure syndromes or myeloproliferative disorders

Recipient Exclusion Criteria:

* Pregnant or lactating women.
* Subjects with other major medical or psychiatric illnesses which the treating physician feels could seriously compromise tolerance to this protocol.
* Subjects with uncontrolled, progressive infections.
* Subjects who are good candidates for long term disease control with standard chemotherapy or radiation or high dose therapy and autologous support.
* Subjects with active central nervous system (CNS) disease.

Donor Inclusion Criteria:

1. Donor must be capable of providing informed consent. If 14-17 years of age, a 'single patient exemption' from the local Institutional Review Board must be obtained.
2. Donor must not have any medical condition which would make mobilization or apheresis more than a minimal risk, and should have the following:

   1. Adequate cardiac function by history and physical examination. Those with a history of cardiac failure or infarction should be evaluated by a cardiologist prior to donation
   2. Adequate hematopoietic function with hematocrit ≥ 30%, white blood cell count of 3000, and platelets 100,000.
3. Females should not be pregnant or lactating and have a negative serum pregnancy test within 1 week of beginning mobilization if of child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2008-02; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rizzieri, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- [Result] Kanda J, Long GD, Gasparetto C, Horwitz ME, Sullivan KM, Chute JP, Morris A, Shafique M, Li Z, Chao NJ, Rizzieri DA. Reduced-intensity allogeneic transplantation using alemtuzumab from HLA-matched related, unrelated, or haploidentical related donors for patients with hematologic malignancies. Biol Blood Marrow Transplant. 2014 Feb;20(2):257-63. doi: 10.1016/j.bbmt.2013.11.010. Epub 2013 Nov 20. PMID 24269380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 170 transplant recipients were recruited through the Adult Bone Marrow Transplant Program at Duke University Medical Center. Recruitment began in February, 2008 and ended in June, 2013. 33 recipients were screen failures. 94 donors were consented for leukapheresis.
Pre-assignment Details: Recipients had history and exam, labs, x-ray, and possible bone marrow aspirate. Radiation therapy may be used prior to transplant for minimal active disease. Donor selection included a 5-6/6 matched sibling as the first choice, a matched unrelated donor as the second choice, or a 3-5/6 partially matched family member as the third choice.
Groups:
- Cohort A - Lymphoid Disease: Non-myeloablative stem cell transplant (SCT): Donor will receive Granulocyte colony-stimulating factor (G-CSF) 8 mcg/kg/d subcutaneously twice daily for 4 days, until pheresis is completed or until white blood cells > 100,000. Recipients will be premedicated with Benadryl 50 mg intravenously (IV) or orally (PO), and acetaminophen 650 mg PO (or hydrocortisone 50-100 mg IV on first day). The preparative regimen is 4 days of daily fludarabine at 40 mg/m2/d infused over 30 minutes; melphalan 140 mg/m2/d for 1 day administered over 15 minutes; 4 days of Alemtuzumab at 20 mg/d in 250 ml of normal saline infused over 3 hours. The PBSCs will be infused over 2-4 days. Participant evaluations will occur 2 times per week by physical exam for toxicity through day 45.
- Cohort B - Myeloid Disease: Non-myeloablative stem cell transplant (SCT): Donor will receive granulocyte colony stimulating factor (G-CSF) 8 mcg/kg/d subcutaneously twice daily for 4 days, until pheresis is completed or until white blood cells > 100,000. Recipients will be premedicated with Benadryl 50 mg intravenously (IV) or orally (PO), and acetaminophen 650 mg PO (or hydrocortisone 50-100 mg IV on first day). The preparative regimen is 4 days of daily fludarabine at 40 mg/m2/d infused over 30 minutes; melphalan 140 mg/m2/d for 1 day administered over 15 minutes; 4 days of Alemtuzumab at 20 mg/d in 250 ml of normal saline infused over 3 hours. The prep regimen will begin on day -5 or day -4 and busulfan 130mg/m2/d for 2 days over 3 hours. The PBSCs will be infused over 2-4 days. Participant evaluations will occur 2 times per week by physical exam for toxicity through day 45.
- Donor: 1. 5-6/6 matched sibling who meets the other donor criteria is the first choice,
  2. Matched Unrelated Donor (MUD) is the second choice*, and
  3. 3-5/6 partially matched family member (if 5/6 then this donor is not a sibling as that would be first choice) is the third choice for donor type.
  Multiple choices for 3-5/6 human leukocyte antigen (HLA) matched family member donors order of choice will be best match, then cytomegalovirus (CMV) negativity, then Killer-cell immunoglobulin-like receptors (KIR) mismatching (for natural killer [NK] cell activity), then history of pregnancy. All subjects without an available matched sibling must have a donor search initiated with the national bank. If potential high resolution matches are found but not utilized, the reason for proceeding with a partially matched family member should be documented (i.e. donor not available, not enough time to allow MUD donor work up and collection due to high risk nature of the subject's disease, etc).
Period: Overall Study
Arm/Group | Cohort A - Lymphoid Disease | Cohort B - Myeloid Disease | Donor
Started | 80 | 57 | 94
Completed | 24 | 11 | 84
Not Completed | 56 | 46 | 10
Not completed — Death | 56 | 46 | 0
Not completed — Recipient death | 0 | 0 | 10

BASELINE CHARACTERISTICS:
Population: Participants who proceeded to therapy and transplant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - Lymphoid Disease | Cohort B - Myeloid Disease | Total
Number analyzed (Participants) | 80 | 57 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 40 | 113
  >=65 years | 7 | 17 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 24 | 59
  Male | 45 | 33 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 70 | 51 | 121
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 80 | 57 | 137
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 80 | 57 | 137

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival
Description: Estimate disease free survival rates in participants treated with an alemtuzumab T cell depleted, reduced intensity preparative regimen followed by allogeneic hematopoietic transplantation. Disease-free survival (DFS), progression-free survival (PFS), and overall survival (OS) rates after SCT were estimated using the Kaplan-Meier method. We performed univariate comparisons by using the log-rank test. DFS was defined as the period of time between the day of transplantation and either disease relapse or death due to the disease. The following variables were considered as confounders: recipient age, recipient sex, disease (myeloid or lymphoid), disease risk (standard or high), and donor type (MRD, MUD, or HAPLO donor). The percentage of participants who were disease free at 2 years is reported by donor type.
Time Frame: 2 years
Population: All subjects with complete response. Cohort A (n=62) had acute or chronic leukemia (ALL or CLL), lymphoma, or myeloma. Cohort B (n=62) had acute or chronic myeloid leukemia (AML or CML), myelodysplastic disorder or myeloproliferative disorder. DFS was analyzed by type of donor (Matched Unrelated Donor; Matched Related Donor; Haplo-identical).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort A & B- Lymphoid & Myeloid Disease: Non-myeloablative Stem Cell Transplant (SCT): Donor will receive Granulocyte colony-stimulating factor (G-CSF) 8 mcg/kg/d subcutaneously twice daily for 4 days, until pheresis is completed or until white blood cells > 100,000. Recipients will be premedicated with Benadryl 50 mg intravenously (IV) or orally (PO), and acetaminophen 650 mg PO (or hydrocortisone 50-100 mg IV on first day). The preparative regimen is 4 days of daily fludarabine at 40 mg/m2/d infused over 30 minutes; melphalan 140 mg/m2/d for 1 day administered over 15 minutes; 4 days of Alemtuzumab at 20 mg/d in 250 ml of normal saline infused over 3 hours. The prep regimen for myeloid disease will begin on day -5 or day -4 and busulfan 130mg/m2/d for 2 days over 3 hours. The Peripheral Blood Stem Cells (PBSCs) will be infused over 2-4 days. Participant evaluations will occur 2 times per week by physical exam for toxicity through day 45.
Arm/Group | Cohort A & B- Lymphoid & Myeloid Disease
Number analyzed (Participants) | 124
percentage of participants
  Matched Related Donors (MRD); n=38 | 47 [29 to 63]
  Matched Unrelated Donors (MUD); n=53 | 23 [12 to 36]
  Haploidentical related (HAPLO) donors; n=33 | 16 [5 to 33]

2. Secondary Outcome: Immune Recovery
Description: Evaluate immune recovery following this reduced intensity allogeneic immunotherapy. Quantification of CD3+, CD4+, and CD8+ T cells was performed by flow cytometry on fresh peripheral blood at approximately 1 month before transplantation and then 1.5, 3, 6, and 12 months after transplantation. The immune recovery rates of the CD3+, CD4+, and CD8+ T cells in the MRD, MUD, and HAPLO groups were compared by performing an analysis of variance at each time point after transplantation. The median T cell counts at 12 months for each type of cell are reported by donor type.
Time Frame: 1 year
Population: All subjects with complete response. Cohort A (n=62) had acute or chronic leukemia (ALL or CLL), lymphoma, or myeloma. Cohort B (n=62) had acute or chronic myeloid leukemia (AML or CML), myelodysplastic disorder or myeloproliferative disorder. Analysis by type of donor (Matched Unrelated Donor; Matched Related Donor; Haplo-identical).
Measure: Mean (Standard Deviation); unit: T cells/μL
Groups:
- Cohort A & B- Lymphoid & Myeloid Disease: Non-myeloablative Stem Cell Transplant (SCT): Donor will receive Granulocyte colony-stimulating factor (G-CSF) 8 mcg/kg/d subcutaneously twice daily for 4 days, until pheresis is completed or until white blood cells > 100,000. Recipients will be premedicated with Benadryl 50 mg intravenously (IV) or orally (PO), and acetaminophen 650 mg PO (or hydrocortisone 50-100 mg IV on first day). The preparative regimen is 4 days of daily fludarabine at 40 mg/m2/d infused over 30 minutes; melphalan 140 mg/m2/d for 1 day administered over 15 minutes; 4 days of Alemtuzumab at 20 mg/d in 250 ml of normal saline infused over 3 hours. The Peripheral Blood Stem Cells (PBSCs) will be infused over 2-4 days. Participant evaluations will occur 2 times per week by physical exam for toxicity through day 45.
Arm/Group | Cohort A & B- Lymphoid & Myeloid Disease
Number analyzed (Participants) | 124
T cells/μL
  Matched Related Donors (MRD) n=38 - CD3+ Tcells/uL | 700 (100)
  Matched Unrelated Donors(MUD) n=53 - CD3+Tcells/uL | 550 (150)
  Haploidentical related (HAPLO) n=33 -CD3+Tcells/uL | 500 (200)
  Matched Related Donors (MRD) n=38 - CD4+ Tcells/uL | 225 (30)
  Matched Unrelated Donors (MUD) n=53 -CD4+Tcells/uL | 140 (20)
  Haploidentical related (HAPLO) n=33 -CD4+Tcells/uL | 150 (55)
  Matched Related Donors (MRD) n=38 - CD8+ Tcells/uL | 420 (100)
  Matched Unrelated Donors (MUD) n=53 -CD8+Tcells/uL | 350 (150)
  Haploidentical related (HAPLO) n=33 -CD8+Tcells/uL | 300 (150)

3. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) rates after stem cell transplant were estimated using the Kaplan-Meier method. We performed univariate comparisons by using the log-rank test. PFS was defined as the period of time between the day of transplantation and either the day underlying disease progression was documented or death occurred by any cause. The following variables were considered as confounders: recipient age, recipient sex, disease (myeloid or lymphoid), disease risk (standard or high), and donor type (MRD, MUD, or HAPLO donor). The percentage of participants progression free at 2 years is reported by donor type. Progression = > 25% increase of serum M-protein and/or urine M-protein. Also, an absolute increase in bone marrow plasma cells > 10%, new bone lesions or soft tissue plasmacytomas or increase in the size of existing bone lesions or soft tissue plasmacytomas or development of hypercalcemia that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: 2 years
Population: All participants who received transplant. Cohort A (n=62) had acute or chronic leukemia (ALL or CLL), lymphoma, or myeloma. Cohort B (n=62) had acute or chronic myeloid leukemia (AML or CML), myelodysplastic disorder or myeloproliferative disorder. Analysis by type of donor (Matched Unrelated Donor; Matched Related Donor; Haplo-identical).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort A & B - Lymphoid & Myeloid Disease: Non-myeloablative Stem Cell Transplant (SCT): Donor will receive Granulocyte colony-stimulating factor (G-CSF) 8 mcg/kg/d subcutaneously twice daily for 4 days, until pheresis is completed or until white blood cells > 100,000. Recipients will be premedicated with Benadryl 50 mg intravenously (IV) or orally (PO), and acetaminophen 650 mg PO (or hydrocortisone 50-100 mg IV on first day). The preparative regimen is 4 days of daily fludarabine at 40 mg/m2/d infused over 30 minutes; melphalan 140 mg/m2/d for 1 day administered over 15 minutes; 4 days of Alemtuzumab at 20 mg/d in 250 ml of normal saline infused over 3 hours. For the myeloid group, the prep regimen will begin on day -5 or day -4 and busulfan 130mg/m2/d for 2 days over 3 hours. The Peripheral Blood Stem Cells (PBSCs) will be infused over 2-4 days. Participant evaluations will occur 2 times per week by physical exam for toxicity through day 45.
Arm/Group | Cohort A & B - Lymphoid & Myeloid Disease
Number analyzed (Participants) | 124
percentage of participants
  Matched Related Donors (MRD) n=38 | 43 [26 to 59]
  Matched Unrelated Donors (MUD) n=53 | 22 [11 to 34]
  Haploidentical related (HAPLO) donor n=33 | 15 [5 to 30]

4. Secondary Outcome: Overall Survival
Description: Estimate overall survival rates in participants treated with an alemtuzumab T cell depleted, reduced intensity preparative regimen followed by allogeneic hematopoietic transplantation. Disease-free survival (DFS), progression-free survival (PFS), and overall survival (OS) rates after SCT were estimated using the Kaplan-Meier method. We performed univariate comparisons by using the log-rank test. OS was defined as the period of time between the day of transplantation and death. The following variables were considered as confounders: recipient age, recipient sex, disease (myeloid or lymphoid), disease risk (standard or high), and donor type (MRD, MUD, or HAPLO donor). The percentage of participants surviving 2 years by donor type is reported.
Time Frame: 2 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort A & B - Lymphoid & Myeloid Disease: Non-myeloablative Stem Cell Transplant (SCT): Donor will receive Granulocyte colony-stimulating factor (G-CSF) 8 mcg/kg/d subcutaneously twice daily for 4 days, until pheresis is completed or until white blood cells > 100,000. Recipients will be premedicated with Benadryl 50 mg intravenously (IV) or orally (PO), and acetaminophen 650 mg PO (or hydrocortisone 50-100 mg IV on first day). The preparative regimen is 4 days of daily fludarabine at 40 mg/m2/d infused over 30 minutes; melphalan 140 mg/m2/d for 1 day administered over 15 minutes; 4 days of Alemtuzumab at 20 mg/d in 250 ml of normal saline infused over 3 hours. The prep regimen for myeloid disease will begin on day -5 or day -4 and busulfan 130mg/m2/d for 2 days over 3 hours. The Peripheral Blood Stem Cells (PBSCs) will be infused over 2-4 days. Participant evaluations will occur 2 times per week by physical exam for toxicity through day 45.
Arm/Group | Cohort A & B - Lymphoid & Myeloid Disease
Number analyzed (Participants) | 124
percentage of participants
  Matched Related Donors (MRD) n=38 | 51 [33 to 66]
  Matched Unrelated Donors (MUD) n=53 | 22 [12 to 35]
  Haploidentical related (HAPLO) donors n=33 | 23 [10 to 39]

5. Other Pre Specified Outcome: Graft Versus Host Disease
Description: Estimate toxicity including graft-versus-host disease (GVHD) in participants treated with an alemtuzumab T cell depleted, reduced intensity preparative regimen followed by allogeneic hematopoietic transplantation. Bone marrow aspiration and/or biopsy were performed 3-5 weeks after transplant to assess donor-cell engraftment. Acute or chronic GVHD was diagnosed and graded according to standard criteria. Toxicity was formally graded using the National Cancer Institute Common Toxicity Criteria version 3.0.
Time Frame: 180 days
Population: All participants who received transplant. Cohort A (n=62) had acute or chronic leukemia (ALL or CLL), lymphoma, or myeloma. Cohort B (n=62) had acute or chronic myeloid leukemia (AML or CML), myelodysplastic disorder or myeloproliferative disorder. Analysis by occurrence of Graft versus Host Disease (GvHD) and Graft Failure and donor type.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort A & B - Lymphoid & Myeloid Disease: Non-myeloablative Stem Cell Transplant (SCT): Donor will receive Granulocyte colony-stimulating factor (G-CSF) 8 mcg/kg/d subcutaneously twice daily for 4 days, until pheresis is completed or until white blood cells > 100,000. Recipients will be premedicated with Benadryl 50 mg intravenously (IV) or orally (PO), and acetaminophen 650 mg PO (or hydrocortisone 50-100 mg IV on first day). The preparative regimen is 4 days of daily fludarabine at 40 mg/m2/d infused over 30 minutes; melphalan 140 mg/m2/d for 1 day administered over 15 minutes; 4 days of Alemtuzumab at 20 mg/d in 250 ml of normal saline infused over 3 hours. The prep regimen for myeloid disease will begin on day -5 or day -4 and busulfan 130mg/m2/d for 2 days over 3 hours.The Peripheral Blood Stem Cells (PBSCs) will be infused over 2-4 days. Participant evaluations will occur 2 times per week by physical exam for toxicity through day 45.
Arm/Group | Cohort A & B - Lymphoid & Myeloid Disease
Number analyzed (Participants) | 124
percentage of participants
  Grade II-IV GvHD (MRD n=38) | 16 [7 to 30]
  Grade II-IV GvHD (MUD n=53) | 26 [14 to 39]
  Grade II-IV GvHD (HAPLO n=33) | 46 [24 to 65]
  Grade III-IV GvHD (MRD n=38) | 3 [0.2 to 12]
  Grade III-IV GvHD (MUD=53) | 13 [5 to 25]
  Grade III-IV GvHD (HAPLO n=33) | 27 [11 to 47]

6. Secondary Outcome: Graft Failure
Description: Estimate toxicity including graft-versus-host disease (GVHD) in participants treated with an alemtuzumab T cell depleted, reduced intensity preparative regimen followed by allogeneic hematopoietic transplantation. Bone marrow aspiration and/or biopsy were performed 3-5 weeks after transplant to assess donor-cell engraftment. Primary Graft Failure was defined as a neutrophil count below 500/μL or the absence of donor-derived hematopoiesis (<5%donor cells) before relapse, death, or re-transplantation. Secondary Graft Failure was defined as the achievement of primary engraftment and a subsequent decrease in neutrophils to 3 consecutive counts of less than 100/μL or the absence of donor-derived hematopoiesis (<5% donor cells) before relapse, death, or re-transplantation.
Time Frame: 180 days
Population: All subjects who received transplant. Cohort A (n=62) had acute or chronic leukemia (ALL or CLL), lymphoma, or myeloma. Cohort B (n=62) had acute or chronic myeloid leukemia (AML or CML), myelodysplastic disorder or myeloproliferative disorder. Analysis by occurrence of Graft versus Host Disease (GvHD) and donor type.
Measure: Number; unit: number of participants
Arm/Group | Cohort A & B - Lymphoid & Myeloid Disease
Number analyzed (Participants) | 124
number of participants
  Graft Failure (MRD n=38) | 1
  Graft Failure (MUD n=53) | 3
  Graft Failure (HAPLO n=33) | 10

ADVERSE EVENTS:
Time Frame: Participants will be evaluated at a minimum of 2 times per week by physical exam for toxicity following Version 3 of the NCI expanded common toxicity criteria through day 45 following the first infusion.
Description: Graft versus Host Disease (GVHD) and other toxicity was graded per NCI's common terminology criteria for adverse events (CTCAE) (3.0).
Groups:
- Cohort A - Lymphoid Disease: Non-myeloablative stem cell transplant (SCT): Donor will receive Granulocyte colony-stimulating factor (G-CSF) 8 mcg/kg/d subcutaneously twice daily for 4 days, until pheresis is completed or until white blood cells > 100,000. Recipients will be premedicated with Benadryl 50 mg intravenously (IV) or orally (PO), and acetaminophen 650 mg PO (or hydrocortisone 50-100 mg IV on first day). The preparative regimen is 4 days of daily fludarabine at 40 mg/m2/d infused over 30 minutes; melphalan 140 mg/m2/d for 1 day administered over 15 minutes; 4 days of Alemtuzumab at 20 mg/d in 250 ml of normal saline infused over 3 hours. The peripheral blood stem cells (PBSCs) will be infused over 2-4 days. Participant evaluations will occur 2 times per week by physical exam for toxicity through day 45.
- Cohort B - Myeloid Disease: Non-myeloablative stem cell transplant (SCT): Donor will receive granulocyte colony stimulating factor (G-CSF) 8 mcg/kg/d subcutaneously twice daily for 4 days, until pheresis is completed or until white blood cells > 100,000. Recipients will be premedicated with Benadryl 50 mg intravenously (IV) or orally (PO), and acetaminophen 650 mg PO (or hydrocortisone 50-100 mg IV on first day). The preparative regimen is 4 days of daily fludarabine at 40 mg/m2/d infused over 30 minutes; melphalan 140 mg/m2/d for 1 day administered over 15 minutes; 4 days of Alemtuzumab at 20 mg/d in 250 ml of normal saline infused over 3 hours. The prep regimen will begin on day -5 or day -4 and busulfan 130mg/m2/d for 2 days over 3 hours. The peripheral blood stem cells (PBSCs) will be infused over 2-4 days. Participant evaluations will occur 2 times per week by physical exam for toxicity through day 45.
Arm/Group | Cohort A - Lymphoid Disease | Cohort B - Myeloid Disease
Serious Adverse Events (participants affected / at risk) | 16/80 | 10/57
Other Adverse Events (participants affected / at risk) | 77/80 | 52/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - Lymphoid Disease (N=80) | Cohort B - Myeloid Disease (N=57)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Death - NOS (General disorders) | 9 (9) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatobiliary/Pancreas (Hepatobiliary disorders) | 1 (1) | 0 (0) — Elevation bilirubin and alkaline phosphate
Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 1 (1) | 1 (2)
Infection - Other (Infections and infestations) | 3 (3) | 3 (3) — Meningitis; Parainfluenza; Herpes Zoster; Nocardia; Sepsis; Hickman line infection; C-Diff
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 2 (2) | 3 (5) — Sepsis; Parainfluenza III; Gram positive cocci (Staph Aureus); Human Herpes Virus 6; Pneumonia; Polyoma virus; Viremia
Infection with grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 2 (3) | 0 (0) — H. pylori; BK virus; Influenza
Infection with unknown ANC (Infections and infestations) | 1 (1) | 0 (0) — Fever possibly due to Human Herpes Virus 6
Altered Mental Status (Nervous system disorders) | 1 (1) | 1 (2)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Death
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Shortness of Breath
CNS - Cerebrovascular Ischemia (Nervous system disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1) — Central Nervous System
Liver dysfunction/failure (Hepatobiliary disorders) | 0 (0) | 1 (1) — Portal hypertension
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - Lymphoid Disease (N=80) | Cohort B - Myeloid Disease (N=57)
Failure to Engraft (Blood and lymphatic system disorders) | 3 (3) | 13 (13)
Diarrhea (Gastrointestinal disorders) | 17 (20) | 4 (4)
Fever without neutropenia (General disorders) | 4 (7) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5)
Mucositis/Stomatitis (Gastrointestinal disorders) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 5 (6) | 3 (3) — Liver laceration; Retroperitoneal bleed; Ulcerative Colitis; Death (4)
Febrile neutropenia (Infections and infestations) | 40 (46) | 22 (23)
Infection - Other (Infections and infestations) | 14 (14) | 4 (5) — Pneumonia; Sepsis; Viremia; Human Herpes Virus 6; Herpes Simplex Virus; Cytomegalovirus; Fungal Pneumonia
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 53 (118) | 41 (90) — Bacteremia; Polyoma; Cytomegalovirus; Viremia; Varicella Zoster; Human Herpes Virus 6; Parainfluenza; Respiratory syncytial virus; Penicillium; Vancomycin-resistant enterococcus; Nocardia; Strep Viridans; Gram+ cocci; Ecoli; C-Diff; Klebsiella; MRSA
Infection with normal ANC or grade 1 or 2 neutrophils (Infections and infestations) | 42 (101) | 18 (37) — Varicella Zoster; Cytomegalovirus; Viremia; Pneumonia; Stenotrophomonas Maltophilin; Herpes Simplex Virus; Human Herpes Virus 6; Gram+ cocci; Polyoma; Respiratory syncytial virus; C-Diff; Rhizopus; Parainfluenza; BK virus; Staph; MRSA; Gram- rod
Infection with unknown ANC (Infections and infestations) | 5 (12) | 1 (1) — Thrush; Polyoma; Gram negative Sepsis; Gram positive cocci; Cytomegalovirus; Human Herpes Virus 6; Parainfluenza
Creatinine (Metabolism and nutrition disorders) | 8 (8) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 1 (2) — Shortness of Breath
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (5)
Renal/Genitourinary - Other (Renal and urinary disorders) | 7 (8) | 2 (3) — Polyoma nephritis; Dysuria; Foscarnet urethritis; Hematuria; Renal Insufficiency; Renal Failure (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes